CLINICAL TRIAL: NCT06393660
Title: Treatment Use of the CliniMACS® CD34 TCR Alpha/Beta to Prepare Cells for an Unlabeled Indication Using an HLA-Compatible Related or Unrelated Donor for Allogenic Transplant
Brief Title: Treatment Use of the CliniMACS® CD34 TCR Alpha/Beta for Allogenic Transplant (Expanded Access Use)
Status: Available | Type: Expanded Access
Sponsor: Victor Aquino (Other)
Responsible Party: Sponsor-Investigator, Victor Aquino, Professor, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Other Study IDs: STU-2024-0185
Record Dates: First submitted 2024-04-09; First posted 2024-05-01 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Transplant-Related Disorder; GVH - Graft Versus Host Reaction
Keywords: TCR Alpha/Beta; CliniMACS

INTERVENTIONS:
Device: CliniMACS® CD34 TCR Alpha/Beta — CliniMACS System uses an automated antibody/magnetic beads column system that allows efficient depletion of TCRαβ and CD19+ cells without relevant loss of cell viability. Hematopoietic stem cells are retained in sufficient numbers to permit engraftment and hematopoietic reconstitution. Humanitarian Exemption IDE approval has been obtained for CD34+ cell selection as a method of T-cell depletion.

SUMMARY:
The protocol is designed to provide access to patients to the Clinimacs® CD34 TCRαβ system to prepare cells for an unlabeled indication using an HLA-compatible related or unrelated donor for allogenic transplant.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplant (HSCT) is the only known curative therapy for a variety of non-malignant and malignant disorders1-4. Only about 25% of patients have an HLA-matched sibling and in about 16-75% (depending on ethnicity), a 10/10 HLA-matched unrelated donor can be identified. Engraftment failure is a dynamic complex process that may occur with this product due to unbalanced depletion of T-cells between recipient and donor, not only due to low number of CD34 cells. The use of mis-matched or haploidentical donors is associated with a higher risk of post-transplant mortality due to the development of severe graft versus host disease, graft failure and the development of infection due to the use of immunosuppression or T cell depletion. A total of 10 patients will be enrolled. The patients will be divided into 2 strata (haploidentical 7, unrelated donor 3).

ELIGIBILITY:
Recipient Inclusion Criteria:

* Age less than 22 years of age
* No available genotypically matched related donor (sibling)
* Availability of a suitable donor and graft source
* Haploidentical related mobilized peripheral blood cells
* 9/10 or 10/10 allele matched (HLA-A, -B, -C, -DRB1, -DQB1) volunteer unrelated donor mobilized peripheral blood cells

Donor Inclusion Criteria:

* Matching as described in the Recipient and Donor Suitability Criteria
* Size and vascular access appropriate by center standard for peripheral blood stem cell (PBSC) collection. Donors with inadequate peripheral access will require placement of an apheresis catheter for collection.
* Must meet appropriate screening/eligibility requirements:

  * Haploidentical matched family members: screened by center health screens and found to be eligible.
  * Unrelated donors: meet suitability criteria to donate PBSC
  * HIV negative
  * Not pregnant or lactating
  * Recipient must not have high-level donor specific anti-HLA antibodies according to institutional practices.
  * Must agree to donate PBSC
  * Must give informed consent

Recipient Suitability:

- Adequate organ functioning as demonstrated by:

* MUGA ≥ 50% or ECHO >30%
* 24-hour Creatinine Clearance or Glofil ≥ 50 ml/min or Serum Creatinine ≤2 times the upper limit of normal
* DLCO > 65% of predicted value. FEV1 >65% of predicted
* AST / ALT ≤ 2.5 and/or Bilirubin ≤ 1.5 times the upper limit of normal
* Pregnancy test negative
* HIV 1 / 2 (HIV screen) negative with a negative qualitative HIV PCR.
* HTLV I negative
* RPR or VDRL negative
* RVP (Respiratory Viral PCR) with a negative result
* Positive hepatitis testing does not make the patient ineligible. Hepatitis results will be evaluated on a case-by-case basis by the transplant physician to determine donor suitability/eligibility.

Donor Suitability:

- Allowed Donor Sources

* Fully matched sibling donors are not allowed.
* Unrelated donors. HLA typing of at least 10 alleles is required. Donor must be matched at 9/10 or 10/10 alleles (HLA-A, -B, -C, -DRB1, -DQB1). Haploidentical matched family members. Minimum match level full haploidentical (at least 5/10; HLA-A, -B, -C, -DRB1, -DQB1 alleles), but use of haploidentical donors with extra matches (e.g., 6, 7, or 8/10) encouraged.
* Cord blood is not allowed as a stem cell source on this IDE.

Recipient and Donor Exclusion Criteria:

* Pregnant or lactating females are ineligible as the risk to unborn children and infants is unknown
* Presence of life-threatening, uncontrolled opportunistic infection (fungal, bacterial, or viral infections). Patients with history of fungal disease during induction therapy may proceed if they have a significant response to antifungal therapy with no or minimal evidence of disease remaining by CT evaluation.
* HIV or HTLV I/II infection

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Medical Center - Dallas, Dallas, Texas, United States